CLINICAL TRIAL: NCT02031874
Title: Immunogenicity of Inactivated Swine H1N1 Vaccine In HIV Infected Children - The Miami Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Vaccine and Gene Therapy Institute, Florida (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Ivan Gonzalez, Assistant Clinical Professor, University of Miami
Other Study IDs: 20090858; 5P30AI073961 (NIH)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: HIV
Keywords: H1N1; HIV; Immunogenecity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen PBMC for future experiments as per results.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Miami Cohort: Measured vaccine response to H1N1 in HIV perinatally infected children

SUMMARY:
Immunosuppressed patients are at increased risk for complications of influenza infection, including secondary pneumonia and are recommended for annual influenza vaccination. Thus, the appearance of a novel subtype of influenza A virus designated as 2009 swine H1N1 virus has added an extra layer of complexity in the immunization regimen in this population. In general, susceptibility to swine H1N1 infection among young population is higher as young adults and children completely lack protective titers. According to the Center for Disease Control (CDC), 70 percent of people hospitalized with H1N1 have been "high risk" cases, including persons 65 years of age or older, or people with compromised immune systems as observed during HIV infection. This has prompted CDC to include HIV infected children to be one of the five groups to be vaccinated with the new H1N1 vaccine (National Center for Immunization). Currently no information exists about the nature of the immune response to the vaccine against H1N1 swine-origin influenza virus (S-OIV) in HIV infected children. It is unknown whether HIV impairs the immunogenicity of the vaccine predisposing this population to infection with S-OIV. Thus, a pilot proposal is being undertaken to study the mechanism of H1N1 vaccine protection in HIV infected children, by investigating the correlation of infection status with seroresponse, duration of response and development of influenza-like illness following vaccine. Additionally we will establish whether we can identify immune signatures by characteristic gene expression patterns correlating with the vaccine immunogenicity that can be predictive of efficacy for "good" and "suboptimal" vaccination regimen. Data generated will be used to initiate a comprehensive study on the immunogenicity of the influenza vaccines in HIV-infected children and youth, which is critically important to address the health care needs of this vulnerable population.

DETAILED DESCRIPTION:
Patients will be recruited from HIV-1 outpatient clinic at the time the novel H1N1 vaccine becomes available. Demographic data will be collected after enrollment including HIV-1 viral load (VL) and CD4 count from last visit, antiretroviral therapy, gender and age. Patients will be asked to document adverse reactions observed during this study such as tenderness, pain, redness, and swelling at the injection site as well as systemic adverse reactions such as headache, malaise, and muscle aches. A subject will be withdrawn from the study if a serious adverse reaction occurs such as allergic reaction to a vaccine component or development with a progressive neurological disorder without definitive diagnosis. Statistical analysis will be performed after the viral load and CD4 counts are resulted from the day 30. The microneutralization assays and the titers will be analyzed post day 7 and 37. If the cohort does not seem to generate adequate responses, the study will be discontinued and no further samples collected.

Vaccination:

Since immunocompromised persons may have a diminished immune response to Influenza A (H1N1) 2009 Monovalent Vaccine, a higher antigen load will be used for this study as recommended by the National Center for Immunization and Respiratory Diseases and Centers for Disease Control and Prevention. All of the patients will be given a 0.5 ml intramuscular doses of A/California/7/2009 H1N1 strain inactivated vaccine in the deltoid muscle; all patients will receive a second dose after 4 weeks. Each vaccine dose will contain 15 µg each of H1N1 monovalent antigen. Patients under the age of 9 will receive the second vaccine as standard of care, while patients 9 and older will receive a second dose as part of this study.

Study Design:

This is a pilot study designed to recruit 72 patients with CD4 counts of ≥200. Patients will be enrolled on a first come first serve basis and will attempt to reach equal numbers in gender. A dose (15 µg) of the vaccine will be administered at day 0 and 30. Blood samples will be collected as in Table 1 (see Below). At each visit, the total maximum amount collected will be 17.5 ml divided in three individual samples: The first sample will be 5 ml for serum separation used in the detection of Hemagglutination inhibition (HI) titers and micro-neutralization (MN) assays. The second sample will be 10 ml processed for viral load, CD4 counts and ELISPOT functional B cell assays. The third sample will be 2.5 ml collected in a Paxgene RNA tube for future microarray testing. Based on the HI titer and MN responses obtained, the patients will be classified into three distinct subgroups: (a) high responders with ≥ 4 fold titer increases compared to baseline, (b) moderate responders with ≥ 2 and < 4 fold increases and (c) low responders with < 2 fold increases. From these subgroups, up to 25 complete patient's samples from the high and low responders will be selected for microarray studies. The microarray will compare readings from all visits. These preliminary data will serve the basis for future humoral and innate immunity gene activation.

Hemagglutination inhibition (HI) and microneutralization (MN) assays will be performed on blood samples collected as described in Table 1. Two individual samples will be collected in each visit, one will be used for serum separation used in the detection of HI titers and the second sample for viral load, CD4 counts, ELISPOT and Microarray testing. Based on the HI and MN titer responses obtained, the patients will be classified into three distinct subgroups: (a) high responders with ≥ 4 fold titer increases compared to baseline, (b) moderate responders with ≥ 2 and < 4 fold increases and (c) low responders with < 2 fold increases. From these subgroups, up to 25 complete samples from the high, moderate and low responders will be selected for viral load and microarray studies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have a positive ELISA with confirm with a western blot after 18 months of age or a positive DNA or RNA PCR

Exclusion Criteria:

* Patients with hypersensitivity to eggs or chicken protein, neomycin, or polymyxin, or life-threatening reaction to previous influenza vaccination will be excluded. Pregnant individuals will be excluded from the study at this time. Patients with a previous episode of Guillain-Barré Syndrome (GBS) in relation to a previous influenza vaccination, will also be excluded. Allergic reactions, including anaphylactic shock

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Perinatally Infected Children
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine immunogenecity to vaccine | 1 month
  The primary objectives of this proposal are:
  1. To determine the immunogenicity after each of the two doses of inactivated swine-origin H1N1 influenza vaccine in HIV-1 infected children by neutralizing antibody titers, including the durability of response.
  2. To determine whether vaccinated subjects are dependent upon T cell help and HIV virus control for intrinsic B cell function by antigen specific ELSIPOT assay.
  3. To determine whether we can generate immune signatures related to H1N1 immunization dosing and schedule in the high and low responders (CD4 counts >200) by a systems biology approach using gene array and multiparametric immune phenotyping.

SECONDARY OUTCOMES:
Measure Antibody Response | 6 months
  Secondary objectives:
  4. Assess the effect of H1N1 vaccine administration on antibody response to seasonal trivalent influenza vaccine (TIV).
  5. Analyze potential impact of gender in the differences in antibody production, B cell stimulation and changes in both viral load and CD4 counts.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan A Gonzalez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States